CLINICAL TRIAL: NCT06890091
Title: Etude de l'Association Entre la Fatigue Ressentie Par Les Patients et Les Effets Secondaires spécifiques Des CART Cells, au Cours du Premier Mois après l'Administration Pour un Lymphome Non Hodgkinien
Brief Title: Study of the Association Between Fatigue Experienced by Patients and the Specific Side Effects of CART Cells, During the First Month After Administration for Non-Hodgkin's Lymphoma
Acronym: CAR-TIGUE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241779
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Fatigue Symptom; Lymphoma Non-Hodgkin; Chimeric Antigen Receptor T-cell Therapy; Adverse Events
Keywords: Fatigue; CAR-T cells; Chimeric antigen receptor; Adverse events; Lymphoma Non-Hodgkin; Nurse practitionners
MeSH Terms: conditions — Fatigue; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults receiving CAR-T Cell treatment for non-Hodgkin's lymphoma
  Interventions: Other: Fatigue assessment

INTERVENTIONS:
Other: Fatigue assessment — Fatigue score measured by the EORTC QLQ-FA 12 fatigue self-assessment scale

SUMMARY:
The incidence of cancer in 2023 is estimated at 433136 cases, according to INCa. Haemopathies account for 12% of these new cases of cancer cases of cancer, and around two-thirds are lymphoid haemopathies, in particular lymphomas. There are many treatments available for lymphoma. However, the arrival in France in 2018 of immunotherapy treatments such as CAR-T Cells have changed the paradigm of treatment options for certain non-Hodgkin's lymphomas. In these treatments can have both short-term and long-term adverse effects and long-term adverse effects. During hospitalisation for the administration of CAR-T Cells, acute side effects include CRS and ICANS. There is also another complication very specific to this treatment that has been observed in patients: cytopenias. This is despite the fact that one of the symptoms frequently mentioned and felt by patients during the first month after month after treatment is fatigue. Despite numerous studies on the prevalence of fatigue, healthcare professionals often underestimate this symptom. Nurses, and in particular the advanced practice nurse have a crucial role to play in assessing fatigue. The EORTC scale QLQ-FA12 is a multidimensional scale which assesses the physical emotional and cognitive dimensions of fatigue. The theory of symptom management, which was developed in 1994 by the California College of Nursing in San Francisco, is a relevant framework for understanding fatigue in patients. This theory places the patient's experience at the centre of care. This holistic approach provides a detailed framework for understanding this symptom. "According to the theoretical model, measuring the symptom is an important step and characterising it is an essential element in better targeting the actions to be taken". Although CAR-T Cell therapy is innovative and allows long-term remissions, it is important to evaluate and understand how patients live with this treatment. To our knowledge, few studies have been carried out on quality of life, particularly regarding fatigue, following the first month of CAR-T Cell administration. The research question we will address in this study is: "Is there an association between the side effects of CAR-T Cell treatment and the state of fatigue in patients receiving this treatment for non-Hodgkin's lymphoma during the first month?"

ELIGIBILITY:
Inclusion Criteria:

* Adult (age> 18year old)
* Person hospitalised for treatment with CAR-T Cells for non-Hodgkin's lymphoma.
* Person able to understand and read the French language.

Exclusion Criteria:

* Patient under legal protection
* Opposition to research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults receiving CAR-T Cell treatment for non-Hodgkin's lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue score | At day 30
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  30 days after CAR-T cell injection

SECONDARY OUTCOMES:
Fatigue score | At inclusion
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  5 days before CAR-T cells injection
Fatigue score | At day 2
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  2 days after CAR-T cells injection
Fatigue score | At day 10
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  2 days after CAR-T cells injection
Fatigue score | At day 21
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  2 days after CAR-T cells injection
Physical Fatigue subscore | At inclusion
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  5 days before CAR-T cells injection
Physical Fatigue subscore | At day 2
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  2 days after CAR-T cells injection
Physical Fatigue subscore | At day 10
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  10 days after CAR-T cells injection
Physical Fatigue subscore | At day 21
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  21 days after CAR-T cells injection
Physical Fatigue subscore | At day 30
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  30 days after CAR-T cells injection
Cognitive Fatigue subscore | At inclusion
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  5 days before CAR-T cells injection
Cognitive Fatigue subscore | At 2 days
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  2 days after CAR-T cells injection
Cognitive Fatigue subscore | At 10 days
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  10 days after CAR-T cells injection
Cognitive Fatigue subscore | At 21 days
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  21 days after CAR-T cells injection
Cognitive Fatigue subscore | At 30 days
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  30 days after CAR-T cells injection
Emotional Fatigue subscore | At inclusion
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  5 days before CAR-T cells injection
Emotional Fatigue subscore | At 2 days
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  2 days after CAR-T cells injection
Emotional Fatigue subscore | At 10 days
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  10 days after CAR-T cells injection
Emotional Fatigue subscore | At 21 days
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  21 days after CAR-T cells injection
Emotional Fatigue subscore | At 30 days
  European Organization for Research and Treatment of Cancer Fatigue Scale. This is a 12 items questionnaire ranging from 0 to 100. Higher scores indicate more severe fatigue.
  30 days after CAR-T cells injection
Occurence of side events | Until one month
Severity of side events | Until one month

IPD SHARING:
Plan to Share IPD: Undecided